CLINICAL TRIAL: NCT06733857
Title: The Environmental Costs of Building Human Muscle - a Comparison of Greenhouse Gas Emissions, Water Use and Land Use Between Plant-Based and Omnivorous Diets Following Sports Nutrition Protein Recommendations for Muscle Mass Accrual
Brief Title: The Environmental Costs of Building Human Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Game Changers Institute (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 41490987
Record Dates: First submitted 2024-12-04; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Greenhouse Gas Emissions; Water Use; Land Use
Keywords: Life cycle assessment; Environmental impact; Plant-based; Protein source; Hypertrophy; Sustainability
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plant-based (Experimental): Participants were to consume a high protein plant-based diet while completing a 10-week exercise program consisting of 5 exercise sessions per week.
  Interventions: Behavioral: VEG2
- Omnivorous (Active Comparator): Participants were to consume a high protein omnivorous diet while completing a 10-week exercise program consisting of 5 exercise sessions per week.
  Interventions: Behavioral: OMNI2

INTERVENTIONS:
Behavioral: VEG2 — Participants were provided with a caloric target to place them in a ∼0 to 10% energy surplus, and a protein target of 2 g·kg bm-1·d-1. Participants were instructed to avoid animal products for ≥6 d per wk, focusing their intake on protein-rich non-animal-derived foods (for example, mycoprotein-containing products, pulses, soy). To facilitate reaching protein intake targets, the research team provided participants with mycoprotein-containing vegan products (∼1-2 products per day) to be used as the main protein source for some meals. This group also received 105-g mycoprotein (46-g protein, 10-g carbohydrate, 13-g fat, 348 kcal), 35-g post-training, and 70-g before bed.
  Arms: Plant-based
Behavioral: OMNI2 — Participants were provided with a caloric target to place them in a ∼0 to 10% energy surplus, and a protein target of 2 g·kg bm-1·d-1. Participants in OMNI2 were instructed to consume an omnivorous diet, focusing their intake on high-quality animal-derived proteins (that is, meat, milk, yogurt, cheese). To facilitate reaching protein intake targets, the research team provided participants with a weekly supply (∼1-2 products per day) of chicken or beef to be used as the main protein source for some meals. This group also received 59-g supplemental milk protein daily (47-g protein, 2-g carbohydrate, <1-g fat, 198 kcal) 19.5-g to drink post-training and 39-g to drink before sleep.
  Arms: Omnivorous

SUMMARY:
Among the general population, it has been established that plant-based diets confer significant environmental benefits (greenhouse gas emissions, land use, and water use) compared to omnivorous diets.

However, sports nutrition recommendations for supporting resistance exercise-induced gains in muscle mass and strength differ substantially from population-level recommendations, especially for protein intake. Therefore the difference in environmental impact between omnivorous and plant-based diets for adults following such recommendations is as yet unknown.

A prior analysis found that a high-protein, non-animal-derived diet can support resistance training-induced gains in muscle mass and strength to the same extent as a protein-matched omnivorous diet. These findings align with previous research showing that, in the context of a high-protein diet, the source of protein - whether animal or plant-based - does not affect the rate of resistance exercise-induced gains in muscle mass and strength.

The present study therefore plans to retrospectively analyze the diet records from previously published research to determine the difference in environmental impact between the high protein animal-free and omnivorous diets.

The findings could highlight the unique difference in environmental impacts between those following high protein plant-based and omnivorous diets.

DETAILED DESCRIPTION:
The development of skeletal muscle mass is associated with improved athletic performance and cardiometabolic health. Resistance exercise training (RET) and dietary protein ingestion are two key anabolic stimuli that, when repeated consistently over time, promote the accrual of skeletal muscle mass. High protein diets, considerably above the United States RDA of 0.8g·kg bm-1·d-1, are therefore often recommended to support RET adaptations, with meta-analyses highlighting protein intakes of ~1.6g·kg bm-1·d-1 for optimal stimulation of skeletal muscle hypertrophy and strength gains. The Academy of Nutrition and Dietetics suggest that intakes beyond this may be optimal under certain circumstances such as short periods of intensified training or when significantly reducing energy intake.

It has been demonstrated that, in the context of a high-protein diet as a whole, both animal and plant-based protein sources lead to similar RET-induced gains in muscle size and strength. However, the difference in environmental impacts of plant and animal-based protein sources has been shown to be substantial. Both the direct processes related to livestock management (for example, methane production by ruminants) and indirect processes through the inefficiency of using crops for animal feed rather than directly for human consumption contribute to substantially higher environmental impacts for animal-based foods relative to plant-based foods.

Such differences have been highlighted by modeling the environmental impact of replacing population-level food intake with plant-based diets. For instance, a systematic review of 34 studies using environmental life cycle assessments found that, compared to omnivorous diets that followed the same dietary guidelines and caloric content, plant-based diets achieved median reductions of 59% for land use, 45% for water use, and 50% for GHG emissions. Other research has found that high income countries shifting towards a plant-based diet would reduce their annual agricultural production emissions by 61%.

However, established sports nutrition recommendations for protein intake to support RET-induced muscular adaptations differ from general population-level intakes. Therefore the difference in environmental impact between omnivorous and plant-based diets for adults following such recommendations is as yet unknown.

The present study therefore aims to compare the environmental impacts of RET-induced gains in lean mass through consumption of a high protein omnivorous diet with a protein-matched plant-based diet. A previously published study assessed the effects of dietary protein source during a 10-week high volume resistance training program, and found a high protein (~2.0g·kg bm-1·d-1), exclusively plant-based diet and a protein-matched mixed diet led to similar increases in lean mass and strength accrual.

During this study, each participant was required to record dietary intake for a minimum of three days a week, allowing for detailed nutritional analyses. By utilizing environmental life cycle assessments and applying findings from previous meta-analyses, the investigators plan to compare the mean dietary intakes of the two groups, extrapolated across the intervention, to assess each diet's impact on greenhouse gas emissions, land use and water use through a comparative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 - 40 years of age.
* Body mass index between 18 and 30.
* Recreationally active.
* Resistance training experienced (have previous performed resistance exercise, and are familiar with the basic movements).

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes) (as this may affect normal protein metabolism).
* Any diagnosed cardiovascular disease or hypertension (to avoid any complications associated with heavy exercise).
* Elevated blood pressure at the time of screening. (An average systolic blood pressure reading of ≥140mmHg over two or more measurements and an average diastolic blood pressure of ≥90mmHg over two or more measurements.)
* Chronic use of any prescribed or over the counter pharmaceuticals (that may modulate muscle protein metabolism).
* A personal or family history of epilepsy, seizures or schizophrenia.
* Allergic to mycoprotein / Quorn, penicillin, or milk.
* Pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Diet-related greenhouse gas emissions - CO2 equivalents | Applied to diet records for the duration of the 10-week intervention
  Diet-related greenhouse gas emissions defined as CO2 equivalents resulting from food production, calculated by applying environmental life cycle assessments of individual foods and food categories to dietary records.
Diet-related land use - hectares | Applied to diet records for the duration of the 10-week intervention
  Diet-related land use defined as agricultural land required for food production and measured in hectares, calculated by applying environmental life cycle assessments of individual foods and food categories to dietary records.
Diet-related water use - cubic meters | Applied to diet records for the duration of the 10-week intervention
  Diet-related water use defined as freshwater required for food production and measured in cubic meters, calculated by applying environmental life cycle assessments of individual foods and food categories to dietary records.

CONTACTS AND LOCATIONS:
Locations (1):
- Game Changers Institute, Laguna Niguel, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A spreadsheet with full food diary entries (redacted) which the environmental analyses will be based on.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: On request, research institutions will be emailed a protected spreadsheet with full food diary entries (redacted) which the environmental analyses will be based on, as well as the study protocol and the statistical analysis plan.

REFERENCES:
- [Background] Monteyne AJ, Coelho MOC, Murton AJ, Abdelrahman DR, Blackwell JR, Koscien CP, Knapp KM, Fulford J, Finnigan TJA, Dirks ML, Stephens FB, Wall BT. Vegan and Omnivorous High Protein Diets Support Comparable Daily Myofibrillar Protein Synthesis Rates and Skeletal Muscle Hypertrophy in Young Adults. J Nutr. 2023 Jun;153(6):1680-1695. doi: 10.1016/j.tjnut.2023.02.023. Epub 2023 Feb 22. PMID 36822394